CLINICAL TRIAL: NCT03851588
Title: Standard Versus Double Dose Dolutegravir in Patients With HIV-associated Tuberculosis: a Phase 2 Non-comparative Randomised Controlled Trial
Brief Title: Standard Versus Double Dose Dolutegravir in Patients With HIV-associated Tuberculosis
Acronym: RADIANT-TB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: Wellcome Trust (Other); Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Principal Investigator, Prof Gary Maartens, Head of Division of Clinical Pharmacology, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIDRI003
Record Dates: First submitted 2019-02-15; First posted 2019-02-22 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-06

CONDITIONS: HIV Infections; Tuberculosis
Keywords: Antiretroviral therapy; Dolutegravir; Rifampicin; Tuberculosis; Drug-drug interaction
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — dolutegravir

STUDY DESIGN:
Intervention Model Description: Parallel assignment of randomised groups with stratification by ART-naïve versus first-line interrupter status
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supplementary dose (Active Comparator): Dolutegravir-lamivudine-tenofovir fixed-dose combination tablet daily with an additional dolutegravir 50 mg dose taken 12 hours later.
  Interventions: Drug: Dolutegravir 50 mg
- Placebo dose (Placebo Comparator): Dolutegravir-lamivudine-tenofovir fixed-dose combination tablet daily with placebo taken 12 hours later.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Dolutegravir-lamivudine-tenofovir fixed-dose combination tablet daily is not given with a supplementary dose of dolutegravir 50 mg.
  Arms: Placebo dose
Drug: Dolutegravir 50 mg — Dolutegravir-lamivudine-tenofovir fixed-dose combination tablet daily is given with a supplementary dose of dolutegravir 50 mg.
  Other Names: Tivicay 50 mg
  Arms: Supplementary dose

SUMMARY:
The investigators propose to conduct a phase 2 randomised (1:1) double-blind placebo-controlled trial of the dolutegravir-lamivudine-tenofovir fixed dose combination tablet daily with an additional 50 mg dose of dolutegravir/matching placebo taken 12 hours later in ART-naïve or fisrt-line interrupted HIV-infected patients on rifampicin-based anti-tuberculosis therapy. The hypothesis is that virologic outcomes with standard dose dolutegravir-based ART will be acceptable in patients on rifampicin-based anti-tuberculosis therapy.

DETAILED DESCRIPTION:
Dolutegravir is being rolled out to replace efavirenz in first-line antiretroviral therapy (ART) in low-middle income countries (LMICs) because it is more effective, better tolerated, and has a considerably higher genetic barrier to resistance.

Tuberculosis is the commonest cause of HIV-related morbidity and mortality in LMICs. Rifampicin, which is a key component of anti-tuberculosis therapy, induces genes that are important in the metabolism and transport of dolutegravir. The resulting drug-drug interaction between dolutegravir and rifampicin significantly reduces dolutegravir exposure, which can be overcome by increasing the dose of dolutegravir to 50 mg 12 hourly.

The additional dose of dolutegravir will be difficult to implement in high burden settings. Furthermore, the additional dolutegravir tablet increases pill burden and costs. If standard dose dolutegravir is shown to be effective in patients with tuberculosis this would sweep away one of the major barriers to its implementation in LMICs. There are three lines of evidence to support studying standard dose dolutegravir in patients with HIV-associated tuberculosis.

First, there are compelling pharmacokinetic and pharmacodynamic data supporting the therapeutic efficacy of lower dolutegravir exposure. Second, the investigators have conducted a drug-drug interaction study of dolutegravir dosed at 50 mg or 100 mg once daily in healthy volunteers with rifampicin. Although, as expected, concomitant rifampicin significantly reduced dolutegravir exposure at both doses, all dolutegravir trough concentrations on rifampicin were above the protein-adjusted 90% inhibitory concentration (PA IC90). Third, exposure to the first-generation integrase inhibitor raltegravir is also significantly reduced with concomitant rifampicin. A phase 2 study in patients with HIV-associated tuberculosis showed that virologic outcomes were similar with standard and double dose raltegravir. It is plausible that findings could be similar with dolutegravir.

The hypothesis is that virologic outcomes with standard dose dolutegravir-based ART will be acceptable in patients on rifampicin-based anti-tuberculosis therapy. If the proportion of participants who achieve virological suppression on standard dose dolutegravir is acceptable, this would pave the way for a phase 3 trial of dolutegravir 50 mg daily versus an appropriate standard of care regimen, like efavirenz-based ART, in patients with HIV-associated tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection as documented by screening plasma HIV-1 RNA >1000 c/mL
* ART-naïve (short-term antiretroviral use for prevention of mother-to-child transmission will be allowed) or
* ART treatment interrupters on ART <6 months prior to interruption or virologically suppressed (<50 copies/mL or LDL) <6 months prior to interruption
* On rifampicin-based therapy for tuberculosis for <3 months
* CD4 counts >100 cells/µL
* Women of child-bearing potential willing to use adequate contraception (defined as either an intrauterine contraceptive device or hormonal contraception as per national guidelines)

Exclusion Criteria:

* Pregnant/breastfeeding
* Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2 (calculated by the Modification of Diet in Renal Disease (MDRD) study)
* Alanine aminotransferase >3 times upper limit of normal (ULN)
* Allergy or intolerance to one of the drugs in regimen
* Concomitant medication known to significantly reduce or increase dolutegravir exposure (except rifampicin)
* Active psychiatric disease or substance abuse
* On treatment for active AIDS-defining condition other than tuberculosis (participants on maintenance therapy may be enrolled)
* Malignancy
* Any other clinical condition that in the opinion of an investigator puts the patient at increased risk of participating in the study.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Maartens, MMed, Principal Investigator — University of Cape Town
Locations (1):
- Khayelitsha Site B/Ubuntu Clinic, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with other organizations or individuals for further research upon a reasonable request to the University of Cape Town PI, provided that certain conditions are met (including but not limited to the ethical standards upheld by HREC that approved the initial study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From the time the final results are published
Access Criteria: Data will be shared with other organizations or individuals for further research upon a reasonable request to the University of Cape Town PI, provided that certain conditions are met (including but not limited to the ethical standards upheld by HREC that approved the initial study.

REFERENCES:
- [Derived] Griesel R, Zhao Y, Simmons B, Omar Z, Wiesner L, Keene CM, Hill AM, Meintjes G, Maartens G. Standard-dose versus double-dose dolutegravir in HIV-associated tuberculosis in South Africa (RADIANT-TB): a phase 2, non-comparative, randomised controlled trial. Lancet HIV. 2023 Jul;10(7):e433-e441. doi: 10.1016/S2352-3018(23)00081-4. Epub 2023 May 22. PMID 37230101
- [Derived] Griesel R, Hill A, Meintjes G, Maartens G. Standard versus double dose dolutegravir in patients with HIV-associated tuberculosis: a phase 2 non-comparative randomised controlled (RADIANT-TB) trial. Wellcome Open Res. 2021 Jan 11;6:1. doi: 10.12688/wellcomeopenres.16473.1. eCollection 2021. PMID 33954265

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supplementary Dose | Placebo Dose
Started | 53 | 55
Completed | 51 | 52
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Supplementary Dose | Placebo Dose | Total
Number analyzed (Participants) | 53 | 55 | 108
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33 [28 to 38] | 37 [33 to 44] | 35 [31 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 34 | 36 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 53 | 55 | 108
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 53 | 55 | 108
HIV-1 RNA log10 Viral Load [Median (Inter-Quartile Range); unit: log10 copies/mL] | 5.1 [4.6 to 5.6] | 5.2 [4.6 to 5.7] | 5.2 [4.6 to 5.7]
CD4 [Median (Inter-Quartile Range); unit: cells/mm3] | 197 [145 to 260] | 183 [145 to 316] | 188 [145 to 316]

OUTCOME MEASURES:

1. Primary Outcome: Virological Suppression at 24 Weeks
Description: Proportion with HIV viral load <50 copies/mL at 24 weeks analysed by modified intention to treat (ITT), which includes all participants who received at least one dose of dolutegravir, and according to the FDA snapshot algorithm.
Time Frame: 24 weeks
Population: mITT population at 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Supplementary Dose | Placebo Dose
Number analyzed (Participants) | 52 | 53
Participants | 43 | 44

2. Secondary Outcome: Virological Suppression at 12 Weeks (Modified ITT)
Description: Proportion with HIV viral load <50 copies/mL at 12 weeks analyzed modified ITT.
Time Frame: 12 weeks
Population: mITT population at 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Supplementary Dose | Placebo Dose
Number analyzed (Participants) | 53 | 55
Participants | 42 | 46

3. Secondary Outcome: Virological Suppression at 24 Weeks (Per Protocol)
Description: Proportion with HIV viral load <50 copies/mL at 24 weeks analyzed per protocol.
Time Frame: 24 weeks
Population: Per protocol population at 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Supplementary Dose | Placebo Dose
Number analyzed (Participants) | 51 | 52
Participants | 43 | 44

4. Secondary Outcome: Virological Suppression at 48 Weeks (Modified ITT)
Description: Proportion with HIV viral load <50 copies/mL at 48 weeks analyzed modified ITT.
Time Frame: 48 weeks
Population: mITT population at 48 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Supplemental Dolutegravir Arm: Dolutegravir-lamivudine-tenofovir fixed-dose combination tablet daily with an additional dolutegravir 50 mg dose taken 12 hours later.
  Dolutegravir 50 mg: Dolutegravir-lamivudine-tenofovir fixed-dose combination tablet daily is given with a supplementary dose of dolutegravir 50 mg.
- Placebo Arm: Dolutegravir-lamivudine-tenofovir fixed-dose combination tablet daily with placebo taken 12 hours later.
  Placebo: Dolutegravir-lamivudine-tenofovir fixed-dose combination tablet daily is not given with a supplementary dose of dolutegravir 50 mg.
Arm/Group | Supplemental Dolutegravir Arm | Placebo Arm
Number analyzed (Participants) | 49 | 52
Participants | 34 | 35

5. Secondary Outcome: Virological Suppression at 48 Weeks (Per Protocol)
Description: Proportion with HIV viral load <50 copies/mL at 48 weeks analyzed per protocol.
Time Frame: 48 weeks
Population: Per protocol population at week 48
Measure: Count of Participants; unit: Participants
Groups:
- Supplemental Dolutegravir Arm Per Protocol at Week 48: Dolutegravir-lamivudine-tenofovir fixed-dose combination tablet daily with an additional dolutegravir 50 mg dose taken 12 hours later.
  Dolutegravir 50 mg: Dolutegravir-lamivudine-tenofovir fixed-dose combination tablet daily is given with a supplementary dose of dolutegravir 50 mg.
- Placebo Arm Per Protocol at Week 48: Dolutegravir-lamivudine-tenofovir fixed-dose combination tablet daily with placebo taken 12 hours later.
  Placebo: Dolutegravir-lamivudine-tenofovir fixed-dose combination tablet daily is not given with a supplementary dose of dolutegravir 50 mg.
Arm/Group | Supplemental Dolutegravir Arm Per Protocol at Week 48 | Placebo Arm Per Protocol at Week 48
Number analyzed (Participants) | 47 | 46
Participants | 34 | 35

6. Secondary Outcome: CD4 Change at 24 Weeks
Description: Change in CD4 count from screening at week 24.
Time Frame: 24 weeks
Population: mITT population
Measure: Median (Inter-Quartile Range); unit: cells/uL
Arm/Group | Supplementary Dose | Placebo Dose
Number analyzed (Participants) | 52 | 53
cells/uL | 111 [89 to 121] | 101 [84 to 114]

7. Secondary Outcome: Dolutegravir Trough Concentrations
Description: Proportion with dolutegravir trough concentrations above the PA IC90 at week 24
Time Frame: 24 weeks
Population: Participants with available dolutegravir trough concentrations at week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Supplementary Dose | Placebo Dose
Number analyzed (Participants) | 33 | 42
Participants | 32 | 34

8. Secondary Outcome: Grade 3 or 4 Adverse Events
Description: Grade 3 or 4 drug-related adverse events will be accessed throughout the trial.
Time Frame: 48 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Supplementary Dose | Placebo Dose
Number analyzed (Participants) | 53 | 55
Participants | 11 | 10

9. Secondary Outcome: Change in Sleep Assessment From Baseline - Any Treatment Emergent Insomnia After Baseline Assessed at 4 Weekly Intervals Until Week 24 and Then Again at Week 48
Description: Insomnia severity index (ISI scored from 0-28. Score categories: 0-7, no clinical significant insomnia; 8-14, sub-threshold insomnia; 15-21, clinical insomnia (moderate severity); 22-28, clinical insomnia (severe). Measures sleep patterns and how this influences daily functioning and quality of life (assessed through 48 weeks). Measure of participants with treatment emergent insomnia from baseline
Time Frame: Through 48 weeks
Population: Safety population with available scores at baseline and with a baseline score <=7
Measure: Count of Participants; unit: Participants
Arm/Group | Supplementary Dose | Placebo Dose
Number analyzed (Participants) | 51 | 52
Participants | 10 | 4

10. Secondary Outcome: Change in Mental Health Assessment From Baseline Through Week 48
Description: Modified MINI screen (MMS) Mental health questionnaire will be assessed by given at baseline, 12 weeks, 24 weeks, and 48 weeks. The questionnaire is standardized and has been based on the mini international neuropsychiatric interview (version 7.0.0). All questions in the questionnaire require a yes/no answer.
  MMS score increased is worsening MMS includes 22 questions answered yes/no; 2 questions related to experiencing a traumatic event were excluded for a 20 point scale.
  MMS was measured at baseline, week 12, and week 24
  Presenting number of participants with increase in MMS of at least 1 point from baseline through 48 weeks.
Time Frame: Through 48 weeks
Population: Safety population (all participants with baseline assessments available).
Measure: Count of Participants; unit: Participants
Arm/Group | Supplementary Dose | Placebo Dose
Number analyzed (Participants) | 53 | 55
Participants | 2 | 4

11. Secondary Outcome: Serious Adverse Events
Description: Document any serious adverse events that occur throughout the trial.
Time Frame: 48 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Supplementary Dose | Placebo Dose
Number analyzed (Participants) | 53 | 55
Participants | 0 | 5

12. Secondary Outcome: Adverse Events Requiring Discontinuation of an ART Drug
Description: Any adverse event that requires discontinuation of any drug in the ART regimen throughout the trial.
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Supplementary Dose | Placebo Dose
Number analyzed (Participants) | 53 | 55
Participants | 0 | 0

13. Secondary Outcome: Antiretroviral Resistance Mutations Testing by Genotypic Resistance Assay in Participants With Virologic Failure
Description: If a viral load is >1000 copies/mL at week 24 or at week 48, or if the viral load was suppressed and then rebounded to >1000 copies/mL, a sample will be taken for resistance testing. Antiretroviral resistance mutations in participants with virologic failure will be assessed by genotypic resistance assay and compared to stored plasma at baseline to distinguish emergent from pre-treatment resistance.
  Any ART resistance mutations in participants with virological failure by week 48.
Time Frame: Through 48 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Supplementary Dose | Placebo Dose
Number analyzed (Participants) | 53 | 55
Participants | 3 | 3

14. Secondary Outcome: Primary Outcome Differences Among ART-naïve Versus First-line Interruption Status
Description: The primary outcome measure (proportion with HIV viral load <50 copies/mL at 24 weeks analysed by modified intention to treat (ITT), which includes all participants who received at least one dose of dolutegravir, and according to the FDA snapshot algorithm) will be stratified by ART-naïve versus first-line interruption status.
Time Frame: 24 weeks
Population: mITT population
Measure: Count of Participants; unit: Participants
Groups:
- ART Naive Supplemental Dolutegravir Arm; First Line ART Interrupted Supplemental Dolutegravir Arm: Dolutegravir-lamivudine-tenofovir fixed-dose combination tablet daily with an additional dolutegravir 50 mg dose taken 12 hours later.
  Dolutegravir 50 mg: Dolutegravir-lamivudine-tenofovir fixed-dose combination tablet daily is given with a supplementary dose of dolutegravir 50 mg.
- ART Naive Placebo Arm; First Line ART Interrupted Placebo Arm: Dolutegravir-lamivudine-tenofovir fixed-dose combination tablet daily with placebo taken 12 hours later.
  Placebo: Dolutegravir-lamivudine-tenofovir fixed-dose combination tablet daily is not given with a supplementary dose of dolutegravir 50 mg.
Arm/Group | ART Naive Supplemental Dolutegravir Arm | ART Naive Placebo Arm | First Line ART Interrupted Supplemental Dolutegravir Arm | First Line ART Interrupted Placebo Arm
Number analyzed (Participants) | 43 | 42 | 9 | 11
Participants | 36 | 36 | 7 | 8

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Supplementary Dose | Placebo Dose
All-Cause Mortality (participants affected / at risk) | 0/53 | 3/55
Serious Adverse Events (participants affected / at risk) | 0/53 | 5/55
Other Adverse Events (participants affected / at risk) | 3/53 | 0/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supplementary Dose (N=53) | Placebo Dose (N=55)
Treatment resistant oesophageal candidiasis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lichenoid rash secondary to TB treatment (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Trauma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Community acquired pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supplementary Dose (N=53) | Placebo Dose (N=55)
Insomnia (Nervous system disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/88/NCT03851588/Prot_SAP_000.pdf